# The effectiveness of group CBT and exercise in management of Major Depressive Disorder: Protocol for a randomized pilot trial

Marianne Hrabok<sup>1</sup>, Mojtaba Y. Safakar<sup>1</sup>, Graham Gaine<sup>2</sup>, Liana Urichuk<sup>1</sup>, Michal Juhas<sup>1</sup>, Reham Shalaby<sup>1</sup>, Pierre Chue<sup>1</sup>, Mark Snaterse<sup>2</sup>, Judith Mason<sup>2</sup>, Kristina Devoulyte<sup>2</sup>, Laura Leclair<sup>2</sup>, Donna Tchida<sup>2</sup>, Jill Kelland<sup>2</sup>, Pam Coulson<sup>2</sup>, Daniella Sosdjan<sup>2</sup>, Jeff Coulombe<sup>2</sup>, Jason Brown<sup>2</sup>, Katherine Hay<sup>2</sup>, Deanna Lesage<sup>2</sup>, Lucey Flichel<sup>2</sup>, Amy Delday<sup>2</sup>, Sherianna Duiker<sup>2</sup>, Shireen Surood<sup>2,3</sup>, Adam Abba-Aji<sup>1</sup>, Vincent I.O. Agyapong<sup>1</sup>

# \*Corresponding author:

Vincent Israel Opoku Agyapong

Department of Psychiatry, Faculty of Medicine and Dentistry, University of Alberta

1E1 Walter Mackenzie Health Sciences Centre (WMC), 8440 112 St NW, Edmonton, AB T6G 2B7 Canada Phone: 1 780 215 7771 Fax: 1 780 743 3896 Email: agyapong@ualberta.ca

**Source of support**: This work was supported by a Pfizer Depression grant (via Department of Psychiatry, University of Alberta) and support was received from Alberta Health Services

Word count: 2865

Number of tables: 2

**Competing Interests Statement**: All authors have nothing to disclose.

Ethical clearance from Health Ethics Research Board of the University of Alberta, approved on 2018-09-07 - Ref. # Pro 00080975

Operational Approval from Alberta Health Services, approved on 2018-09-12 – Ref. AHS # 43638 Trial registration number on ClinicalTrials.gov: NCT03731728; Pre-results

Version: 2019-03-26

<sup>&</sup>lt;sup>1</sup>Department of Psychiatry, Faculty of Medicine and Dentistry, University of Alberta, Edmonton, Alberta, Canada

<sup>&</sup>lt;sup>2</sup>Addiction and Mental Health, Alberta Health Services, Edmonton, Alberta, Canada

<sup>&</sup>lt;sup>3</sup>Faculty of Social Work, University of Calgary, Calgary, AB, Canada

#### **ABSTRACT**

**Introduction**: Despite evidence in scientific literature indicating the effectiveness of both Cognitive-Behavior Therapy (CBT) and physical exercise in the management of Major Depressive Disorder (MDD), few studies have directly compared them.

**Objective**: This study will evaluate and compare the effectiveness of group CBT versus physical exercise versus only wait-listing to receive treatment as usual (TAU) in the management of MDD. The investigators hypothesize that participants with MDD assigned to the group CBT or exercise arms of the study will achieve superior outcomes compared to participants wait-listed to receive TAU only.

Methods and analysis: This prospective rater-blinded randomized controlled trial assesses the benefits of group CBT and exercise for participants with MDD. 120 patients with MDD referred to Addiction and Mental Health clinics in Edmonton will be randomly assigned to one of the three equal-size arms of the study to receive either weekly sessions of group CBT plus TAU or group exercise 3 times a week plus TAU or only TAU for 14 weeks. Participants will be assessed at enrollment, three and six months post enrolment, mid-treatment, and at treatment completion for primary (functional and symptom variables) and secondary outcomes (service variables and healthcare utilization). In addition, participants in the intervention groups would be evaluated weekly with one functional measure. The data will be analyzed using repeated measures and effect size analyses, and correlational analyses will be completed between measures at each time point.

**Ethics and dissemination**: The study will be conducted in accordance with the Declaration of Helsinki (Hong Kong Amendment) and Good Clinical Practice (Canadian Guidelines). Written informed consent will be obtained from each subject. The study has received ethical clearance from Health Ethics Research Board of the University of Alberta (Pro 00080975), operational approval from the provincial health authority (AHS 43638) and is registered with clinicaltrials.gov. The results will be disseminated at several levels, including patients, practitioners, academics/researchers, and healthcare organizations.

Trial registration number on ClinicalTrials.gov: NCT03731728; Pre-results.

**Keywords**: depression, Major Depressive Disorder, cognitive behavior therapy, group CBT, exercise.

# Strengths of this study

- Randomization of participants will ensure that patients in the three treatment arms have fairly similar psychiatric morbidity at baseline
- Blinding of outcome assessors and the use of self-rating scales for the primary outcome measures will ensure the elimination of bias in outcome measures.

# Limitation of this study

 The rather small sample size may reduce the study power which will limit the ability of the study to detect differences in outcome measures between participants in the three treatment arms

# INTRODUCTION

# **Background** and rationale

Depressive disorders are a major public health problem. For example, the global prevalence of depressive disorders is over 4%, and depression is the single largest contributor to non-fatal health loss [1]. There is a need to identify interventions that are relatively cost-efficient, scalable, and can be offered to many people. Treatment for depressive disorders typically includes anti-depressant medication and/or counselling and psychotherapy.

Exercise as a form of treatment for depressive disorders, especially of mild-to-moderate severity, has evidence of benefit [2, 3, 4, 5]. In fact, the magnitude of the effect of exercise as a treatment for depression is reported to be comparable to conventional treatment [6, 7]. An umbrella review of systematic reviews and meta-analyses of the use of exercise to treat depressive symptoms in older adults, for example, concluded that "exercise is safe and efficacious in reducing depressive symptoms in older people" and exercise "should be considered as a core intervention in the multidisciplinary treatment of older adults experiencing depression" [8]. A meta-analysis adjusting for publication bias, concluded that "exercise has a large and significant antidepressant effect in people with depression" [9]. The mechanisms by which exercise decreases depressive symptoms may include biological mechanisms, such as anti-inflammatory effects [10] or increasing neurotransmitter levels implicated in depression [11]. Other mechanisms may include increase in self-efficacy [10] or enhanced social interaction [12].

Despite this strong evidence base, few studies have incorporated multiple treatment conditions in a randomized controlled trial design, and few studies appear to have assessed the effect of group CBT in comparison to exercise. A randomized clinical trial that assigned 54 mild to moderately depressed patients to a combined CBT plus exercise condition vs. a CBT only condition [13] found superior outcomes in suicidal ideation, depression, and activities of daily living in the combined condition compared to group CBT only. However, few studies could be found that compared group CBT, group exercise, and wait-listing for treatment as usual conditions. This is important in further delineating the effective components of treatment for mild to moderate depression, and results have implications for service delivery and clinical recommendations in the treatment of depression within healthcare organizations in Alberta and beyond. Specifically, patients with MDD referred to Addiction and Mental Health Clinics in Edmonton Zone may wait for weeks before receiving individual treatment. Thus, group treatment conditions examined in this study may serve as an expedient treatment avenue to decrease wait-list times for patients with MDD and improve outcomes.

# **Aim and Objectives**

The aim of the project is to conduct a randomized pilot trial to evaluate the feasibility and effectiveness of group CBT and group exercise on depression symptom scores and functioning. The client outcomes will be organized according to: functional variables (relationships, well-being, physical activity), symptom variables (change in depressive symptoms scores), and service variables (patient compliance, retention in treatment, patient satisfaction).

Given the aim, one objective of the project are to compare mean changes in functioning, clinical symptoms, and service satisfaction variables from enrolment baseline to 12 weeks post enrolment for:

1) participants receiving group CBT plus wait-listed to receive TAU; 2) participants receiving scheduled exercise plus wait-listed to receive TAU; and 3) participants only wait-listed to receive TAU. Another objective of the study is to compare mean changes in functioning, clinical

symptoms, and service satisfaction variables from treatment baseline to 7 and 14 weeks post-treatment commencement for: 1) participants receiving group CBT plus wait-listed to receive TAU and 2) participants receiving scheduled exercise plus wait-listed to receive TAU.

# **Hypothesis**

The investigators hypothesize that participants enrolled in the group CBT or group exercise treatments while wait-listed to receive TAU will achieve statistically superior outcomes at 12 weeks post enrollment compared to participants only wait-listed to receive TAU on each outcome measure used. We expect that participants enrolled in group CBT plus TAU will have comparable outcomes to those enrolled in the group exercise plus TAU arm of the study at 7and 14 weeks post treatment commencement.

# MATERIALS AND METHODS

# Overview of study design, timeline and participant selection

This study will be a longitudinal, prospective, parallel design, three-arm, rater-blinded randomized clinical trial with a recruitment period of six months and an observation period of 14 weeks (plus waiting time) for each participant. The study will be executed according to the timelines specified in the Gantt chart in Table1.

The research will be carried out in a municipal recreational centre as well as Addiction and Mental Health clinics in Edmonton, a large, socio-demographically diverse city in Western Canada [14]. Potential participants will be recruited from the Addiction and Mental Health Intake Clinic in Edmonton. Patients with depression at intake assessment who are presumed to meet the inclusion criteria of the study will be invited to enroll.

To confirm the diagnosis of MDD using DSM-5 criteria, potential participants will be sent to the Mood and Anxiety clinic or Urgent Clinics in Edmonton where they will be assessed by one of a group of psychiatrists or psychiatry residents who are independent from the study team. The psychiatrist or resident may or may not initiate, continue or adjust pharmacotherapy. The diagnosis will be communicated to the study coordinator and clinic nurse. The participants with MDD will be informed of their eligibility to participate in the study and will be considered for randomization after providing informed consent whereas patients with other diagnoses will be informed of their exclusion from the study and will be directed to receive an appropriate treatment for their condition.

After diagnostic confirmation by a psychiatrist, a research assistant who is trained in study procedures will provide the potential participants with an information leaflet about the study and answer any related questions they may have. All potential participants who agree to take part in the study will provide written informed consent prior the completion of baseline assessment measures and randomization.

Patients who are 18 to 65 years of age, have been referred by a primary care provider or self-referred to the Addiction and Mental Health Intake Clinic in Edmonton, have received a primary diagnosis of MDD from a consultant psychiatrist based on DSM-5 criteria, and have provided written informed consent will be included in the study. Patients will be ineligible if they do not meet the above inclusion criteria, have not provided informed consent, or have a diagnosis of Bipolar Disorder, Schizophrenia or Schizoaffective Disorder.

At baseline, demographic and contact information will be collected. The participant's name and contact information will be collected only for use in future communication or for arrangement of treatment, assessment and follow-up sessions.

Participant's Medical Record will also be reviewed at two points, at enrolment and 6 months after enrolment, to gather information about the participant's use of health services in the past 6 months and compare service utilization among the groups and determine if participation in the intervention groups impacts the use of other health services in the short term. This same data can also be used for any economic analyses (i.e., cost-effectiveness) that will be conducted. All the data will be stored for a minimum of 7 years prior to destruction as per the research ethics board requirements, and research ethics board requirements pertaining to collection and storage of information will be followed.

Table 1: Gantt chart for group CBT and exercise project

| | | Year 1 Start Date-End Date | | | | Year 2 Start Date-End Date | |
|---|---|---|---|---|---|---|---|
| Milestone No. | Milestones | Q1 | Q2 | Q3 | Q4 | Q1 | Q2 |
| Milestone 1: Setting up of infrastructure for group CBT and gymnasium | | | | | | | |
| 1.1 | Assembling of group CBT facilitators and setting of gymnasium in the community | | | | | | |
| Milestone 2: The recre | uitment of study participants | | | | | | |
| 2.1 | Recruitment, baseline assessment, randomization | | | | | | |
| 2.2 | Assignment into one of the three arms of the study | | | | | | |
| 2.3 | Delivery of group CBT, exercise, and/or TAU to participants | | | | | | |
| Milestone 3: Follow-u | p assessment of study participants | | | | | | |
| 3.1 | Follow-up assessments of individual study participants (Excluding satisfaction surveys) | | | | | | |
| 3.2 | Follow-up satisfaction survey of participants all groups | | | | | | |
| Milestone 4: Data com | npilation, analysis and preparation of rep | oorts, p | ublicati | ons and | presenta | tions | |
| 4.1 | Data compilation | | | | | | |
| 4.2 | Data Analysis | | | | | | |
| 4.3 | Preparation of reports, publications and presentations | | | | | | |

#### **Interventions**

Participants enrolled in the group CBT plus TAU condition will be wait-listed to receive TAU and will receive a 2-hour session of group CBT every week for 14 weeks. Participants enrolled in the group exercise plus TAU arm of the study will be wait-listed for TAU and will receive 50 minutes of scheduled and facilitated exercises three times a week for 14 weeks. Participants in the TAU only arm of the study will be wait-listed to receive individual therapy or counselling from a therapist as per current standard protocol for managing patients with MDD in Addiction and Mental Health Clinics in Edmonton Zone. All above participants may or may not receive pharmacotherapy as prescribed by a psychiatrist who is independent from the study team.

Group CBT: The group CBT will be offered in Addiction and Mental Health Clinics of Edmonton at 3 clinics: Edmonton Community Mental Health Clinic, Edmonton Hope and Wellness Centre, and AHS Clinical Psychology Service. All therapists will use a manualized CBT protocol with the same handouts and schedule developed based on the book "Mind Over Mood". It will be provided to a group of maximum 10 participants. Each session will be 2 hours long and will be provided by certified therapists with special training to deliver group CBT. The structure of the session will be agenda setting, check-in, review of homework, new concepts/skills, homework assignment, and feedback.

**Group exercise**: For scheduled group exercise, the research team will follow the current recommendations based on a literature review for the use of exercise for the treatment of depression, as well as Canadian Physical Activity Guide recommendations. Scheduled group exercises incorporate the following parameters:

Type – aerobic or strength training exercises

Dose -3 times per week

Intensity- moderate [participant self-rated physical activity of a 6 or 7 on the Borg Perceived Exertion (BPE) scale of 10, relative to the individual's personal capacity]. Moderate heart rate level will be calculated (65% to 75 % of maximum heart rate) for each participate at the beginning of the study and they will have access to heart rate monitors to gain an understanding of what moderate intensity feels like in their body

Time -50 minutes in moderate heart rate zone) per session with 3 sessions per week (150 minutes/week).

Duration – 14 weeks

Other - with supervision: Physical exercise sessions will be run by CanFit Pro or AFLCA certified Recreational Therapists who will assess safety of patients' involvement in physical activity using "Par-Q & You" questionnaire before initiation of the study and address any physical problems to minimize the risk of any adverse events happening during sessions. This form is a screening tool to determine safe participation in exercise. Participants identified as potentially at risk with physical activity will require clearance to participate by his/her medical doctor.

Participants will have an opportunity to choose from a variety of physical activities in order to facilitate a meaningful physical activity experience which is important for long term maintenance. Participants will have the opportunity to engage in three of the following fitness programs per week for fourteen weeks: Monday: Individual fitness for 50 minutes; Tuesday: Group exercise or individual fitness for 50 minutes; Wednesday: Aqua/swimming for 50 minutes; Thursday: Walking track and group exercise for 50 minutes; Friday: Pole walking or hiking according the season for 50 minutes

All participants must consent to participate in the study facilitated exercise groups to be considered in the study because supervision and guidance is required for safety and ensuring

consistent results. During the trial participants are encouraged to participate in the exercise options offered. If the participant engages in the exercise independently it will not be counted as one of their sessions. Once the trial is completed they will be supported to continue exercise options in the community. Participants will be provided with fitness passes and equipment as needed. It will be explained to the participant that although the expense of the equipment is subsidized by the study team to facilitate their participation, they do not have to participate because of this supportive act. They may keep the equipment should they decide to withdraw from the study at any point.

For each session, two Recreation Therapists will provide programming to a maximum of 20 participants. During the sessions the Recreation Therapists will provide participants with information regarding health, wellness, fitness training and understanding exertion levels within exercise. Participants will be encouraged to participate at a moderate level of perceived exertion for the best results (6 to 7 on a 10-point scale). While engaging in the exercise programs the participants will be self-reporting intensity using a rating of perceived exertion scale to the facilitators. Each participant must attend at least 75% of programs (32 sessions out of 42 sessions) during the 14-week period to be considered as having completed the program and for data analysis purposes.

# Sample Size

As this is a pilot study, the research will utilize data that can be elicited from participants who can be enrolled within existing operational resources and time frames. The study will therefore be limited to a sample size of 120, with about 40 patients recruited into each arm of the study.

# **Outcome Measures:**

Outcome measures are detailed in Table 2. Primary outcomes include functional variables (relationships, well-being, physical activity) and symptom variables (depression, risk). Secondary client outcomes include service variables (satisfaction, health utilization).

**Table 2 Outcome Measures** 

| | Construct | Tool | Rater | Time<br>Required | Time Points Assessed | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | At<br>Enrollment | At<br>Start of<br>group CBT<br>or Exercise | 12 weeks<br>Post<br>enrolment | Weekly*<br>during<br>group CBT<br>or<br>Exercise | 7weeks<br>after start<br>of<br>group CBT<br>or<br>Exercise | 14weeks<br>after start<br>of<br>group<br>CBT or<br>Exercise | 6 months<br>after<br>enrollment |
| Symptom<br>Variables | Depressive<br>symptoms | Beck<br>Depression<br>Inventory<br>(BDI-II) [15] | Client | 5 min | Х | Х | Х | | Х | Х | Х |
| | Symptoms,<br>risk level | CORE OM<br>(Symptoms<br>and Risk<br>subscales) | Client | | | | | | | | |
| Functional<br>variables | Inter- personal functioning | CORE OM<br>(Functionin<br>g subscale) | Client | 10 min<br>for 34-<br>items of<br>CORE<br>OM | Х | X | Х | | X | Х | х |
| | Well-being | CORE OM<br>(Well-being<br>subscale) | Client | | | | | | | | |
| | Physical<br>Activity | Internationa<br>I Physical<br>Activity<br>Questionnai<br>re | Client | 5 min | Х | Х | | | Х | Х | |
| Symptom<br>and<br>functional<br>variables | Symptoms,<br>risk,<br>interpersonal<br>functioning<br>and wellbeing | CORE-10<br>OM | Client | 5 min | | | | Х | | | |
| Service<br>variables | Patient<br>Satisfaction<br>with Service | Addiction<br>and Mental<br>Health<br>Client<br>Experience<br>Survey | Client | 5 min | | | | | X | X | |
| | Health<br>Utilization | Data<br>extraction | Research<br>Team | - | Х | | | | | | Х |
| Total Time for participant | | | | | 20 min | | | 25 min | 25 min | | |

<sup>\*</sup>Except week 7 and 14 when CORE 34 OM will be administered

# **Randomization and Blinding**

Randomization will be enacted via randomly generated codes. Each study participant will receive a randomization code. Because it will not be possible for participants to be blinded, treatment allocation will be made explicit to them as soon as randomization is concluded. Outcome assessors will be blinded to treatment group allocation by not involving them in discussions about study participants and not granting them access to the database that contains the randomization code. In addition, study participants will self-complete all outcome assessments with the assessor facilitating procedural aspects if needed. Moreover, these assessors will not be involved in data analysis. After data collection is complete all data will undergo a blind review for the purposes of finalizing the planned analysis.

# Follow-up Assessment

12 and 24 weeks after baseline assessments, a blinded researcher will contact study participants in all three arms of the study and assist them in the completion of a range of assessment tools related to the outcome measures. The number of treatment sessions (group CBT, group exercise or individual therapy) participants have received at each time point would be recorded for participants in all treatment arms. In addition, participants in the group CBT and exercise arms of the study would complete assessments tools weekly during the sessions and also at mid-treatment (7 weeks after starting treatment) and at the end of the treatment (14 weeks after the treatment commencement). These self-rated assessments would be coordinated by the group facilitators.

# **Statistical Methods**

The primary goal of the statistical analysis will be to produce summary descriptive statistics for the longitudinal data, which will provide estimates for future sample size calculations and enable calculation of effect size. For the three arm trial, we will compare mean change scores for primary and secondary outcome measures from enrolment baseline to 12 weeks and 24 weeks post-enrolment into the study, whilst for the two arm trial, we will compare mean changes scores for primary and secondary outcome measures from treatment baseline to 7 and 14 weeks post-enrolment into treatment in addition to comparing trends in weekly change scores on the CORE-10 OM between the two intervention groups. The data will be analyzed using repeated measures and effect size analyses, and correlational analyses will be completed between measures at each time point. The results of this study will guide the design for a future, more highly powered, study.

# Patient and public involvement

The study was designed and finalized based on feedback from patient representatives. This randomized trial also offers patients the opportunity to provide feedback via the patient satisfaction survey.

#### ETHICS AND DISSEMINATION

The study will be conducted in accordance with the Declaration of Helsinki (Hong Kong Amendment) and Good Clinical Practice (Canadian Guidelines). Written informed consent will be obtained from each participant. The study has received ethical clearance from Health Ethics Research Board of the University of Alberta (Ref. # Pro 00080975) and operational approval from the regional health authority (AHS # 43638). The study is registered with clinicaltrials.gov:

(registration number NCT03731728; pre-result). The results will be disseminated at several levels, including patients, practitioners, academics/researchers, and healthcare organizations.

The investigators team will plan an organizational engagement strategy to advance discussions about feasibility and effectiveness prior to the conclusion of the trial. This will help ensure the findings are a relevant part of decision-making processes in a way that is aligned with study findings as they emerge. This may facilitate planning of a larger study that is endorsed at both leadership and operational levels, so that the potential benefits of the interventions can reach patients in a more timely fashion.

# **DISCUSSION**

The results of the study will provide important information about the effectiveness of group CBT and/or group exercise in treatment of MDD. This will augment the literature in this area, and also provide practical benefits in examining if benefit can be derived from the addition group treatment modalities to TAU. Currently, patients with MDD referred to Addiction and Mental Health Clinics in Edmonton Zone may wait for weeks before receiving care from a health care professional in a one-to-one setting. Long wait may negatively impact patients' well-being, personal and occupational function as well as their satisfaction with care, and a group-based treatment may serve as an alternative for patients with MDD that can be more expediently accessed.

The results of the pilot trial may inform the implementation of a multi-center clinical trial and provide useful information for administrators and clinicians who are interested in incorporating these interventions into existing care. The investigators expect that the pilot findings will inform and support administrative decision-making with respect to further scaling and studying the intervention within the province of Alberta and beyond.

**Authors' Contributions**: The study was conceived and designed by VIOA who also contributed to drafting of the initial and final drafts of the manuscript. MH, MYS, GG and LU contributed to the study design and drafting of the initial and final drafts of the manuscript. PC, MS, JM, KD, LL, DT, JK, PC, DS, JC, JB, KH, DL, LF, AD, SD SS and AAA contributed to the study design and revising the initial draft of the of the manuscript. All authors approved of the final draft of the manuscript prior to submission.

**Acknowledgment**: The study team thank Cathy McAlear for her initial contribution to the exercise component of the trial design

**Funding Statement**: This work was supported by a Pfizer Depression grant (via Department of Psychiatry, University of Alberta) and support was received from Alberta Health Services.

**Competing Interests Statement**: All authors have nothing to disclose.

#### References

- 1. World Health Organization. Depression and other common mental disorders: global health estimates. 2017 Licence: CC BY-NC-SA 3.0 IGO URL: http://apps.who.int/iris/bitstream/handle/10665/254610/WHO-MSD-MER-2017.2-eng.pdf
- 2. Bridle C, Spanjers K, Patel S, Atherton N M, Lamb S E. Effect of exercise on depression severity in older people: systematic review and meta-analysis of randomised controlled trials. The British Journal of Psychiatry. 2012; 201(3), 180–185. <a href="https://doi.org/10.1192/bjp.bp.111.095174">https://doi.org/10.1192/bjp.bp.111.095174</a> PubMed ID: 22945926
- 3. Heinzel S, Lawrence J B, Kallies G, Rapp M A, Heissel A. Using Exercise to Fight Depression in Older Adults: A Systematic Review and Meta-Analysis. 2015; GeroPsych, 28(4), 149–162. https://doi.org/10.1024/1662-9647/a000133
- 4. Josefsson T, Lindwall M, Archer T. Physical exercise intervention in depressive disorders: Meta-analysis and systematic review: Exercise intervention in depressive disorders. Scandinavian Journal of Medicine & Science in Sports. 2014; 24(2), 259–272. <a href="https://doi.org/10.1111/sms.12050">https://doi.org/10.1111/sms.12050</a> PubMed ID: 23362828
- 5. Gill A, Womack R, Safranek S. Does exercise alleviate symptoms of depression? Clinical Inquiries, 2010 (MU), PubMed ID: 20824231
- 6. Cooney G M, Dwan K, Greig C A, Lawlor D A, Rimer J, Waugh F R, Mead G E. Exercise for depression. The Cochrane Database of Systematic Reviews. 2013; (9), CD004366. https://doi.org/10.1002/14651858.CD004366.pub6 PubMed ID: 24938566
- 7. Mead G E, Morley W, Campbell P, Greig C A, McMurdo M, Lawlor D A. Exercise for depression. The Cochrane Database of Systematic Reviews. 2009; (3), CD004366. https://doi.org/10.1002/14651858.CD004366.pub4 PubMed ID: 19588354
- 8. Catalan-Matamoros D, Gomez-Conesa A, Stubbs B, Vancampfort D. Exercise improves depressive symptoms in older adults: An umbrella review of systematic reviews and meta-analyses. Psychiatry Research. 2016; 244, 202–209. <a href="https://doi.org/10.1016/j.psychres.2016.07.028">https://doi.org/10.1016/j.psychres.2016.07.028</a> PubMed ID: 27494042
- 9. Schuch F B, Vancampfort D, Richards J, Rosenbaum S, Ward P B, Stubbs B. Exercise as a treatment for depression: A meta-analysis adjusting for publication bias. Journal of Psychiatric Research. 2016; 77, 42–51. <a href="https://doi.org/10.1016/j.jpsychires.2016.02.023">https://doi.org/10.1016/j.jpsychires.2016.02.023</a> PubMed ID: 26978184
- 10. Euteneuer F, Dannehl K, del Rey A, Engler H, Schedlowski M, Rief W. Immunological effects of behavioral activation with exercise in major depression: an exploratory randomized controlled trial. Translational Psychiatry. 2017; 7(5), e1132. https://doi.org/10.1038/tp.2017.76 PubMed ID: 28509904
- 11. Craft L L, Perna F M. The Benefits of Exercise for the Clinically Depressed. Primary Care Companion to The Journal of Clinical Psychiatry. 2004; 6(3), 104–111, PubMed ID: 15361924
- 12. Huang T T, Liu C B, Tsai Y H, Chin Y F, Wong C H. Physical fitness exercise versus cognitive behavior therapy on reducing the depressive symptoms among community-dwelling elderly adults: A randomized controlled trial. International Journal of Nursing Studies. 2015; 52(10), 1542–1552. https://doi.org/10.1016/j.ijnurstu.2015.05.013 PubMed ID: 26105535
- 13. Abdollahi A, LeBouthillier D M, Najafi M, Asmundson G J G, Hosseinian S, Shahidi S, Jalili M. Effect of exercise augmentation of cognitive behavioural therapy for the treatment of suicidal ideation and depression. Journal of Affective Disorders. 2017; 219, 58–63. https://doi.org/10.1016/j.jad.2017.05.012 PubMed ID: 28525821
- 14. City of Edmonton. 2016 Municipal Census Results. 2017, Sept 14; from https://www.edmonton.ca/city\_government/facts\_figures/municipal-census-results.aspx
- 15. Beck AT, Steer R A, Brown G K. Manual for the Beck Depression Inventory-II. San Antonio, TX: Psychological Corporation. 1996, ISBN-10: 0158018389, ISBN-13: 978-0158018386